CLINICAL TRIAL: NCT00715338
Title: Effects of Oxygen on Lung Tissue During Anesthesia
Status: Terminated | Type: Observational
Why Stopped: poor enrollment
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, John Allan Barwis, Asssistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 70808
Record Dates: First submitted 2008-07-10; First posted 2008-07-15 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Lung Injury, Acute
Keywords: Exhaled Breath Condensate; elective surgery; mechanical ventilation; Isofurans; thrombomodulin; requiring; mechanical; ventilation
MeSH Terms: conditions — Acute Lung Injury; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Collect exhaled breath condensates from patients scheduled for a routine surgical procedure before, during, and after surgery for measurements of IsoFs

Draw blood from patients scheduled for a routine surgical procedure before, during, and after surgery for measurements of serum thrombomodulin.

DETAILED DESCRIPTION:
High concentrations of oxygen are routinely administered to patients undergoing routine surgical procedures even though it is highly likely, at least in patients with normal lung function, that this is unnecessary and in fact may be doing unnecessary harm. Therefore, we plan to assess whether there is any evidence of lung injury during surgery resulted from administration of high concentrations of oxygen by measuring Isofurans (IsoFs) in exhaled breath condensate. In our studies in mice that were exposed to high concentrations of oxygen we also found that circulating levels of thrombomodulin were increased. Thrombomodulin is present in endothelial cells and upon injury they release thrombomodulin into the circulation. Endothelial cell injury is known to occur in hyperoxic-induced lung injury. Therefore, in addition to measuring IsoFs in exhaled breath condensate we will also measure plasma concentrations of thrombomodulin as an indicator of endothelial injury.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class I-III.
* Patient is undergoing elective surgery requiring mechanical ventilation
* Patient is an adult, 18 - 80 years old.
* Subject has voluntarily signed and dated the informed consent document approved by the Institutional Review Board (IRB).

Exclusion Criteria:

* Surgical procedures boarded for less than 2 hours
* Current Smoker
* All Cardiac, Thoracic and/or Vascular surgeries involving the chest
* Patient unable to cooperate.
* Chronic airway diseases
* Asthma
* Medical contraindication to anesthetic technique (allergy, cardiac condition, neurologic condition, localized infection, bleeding disorder).
* Subjects who are pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for a routine surgical procedure
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Barwise, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt University Medical Center Department of Anesthesiology — http://www.vandydreamteam.com